CLINICAL TRIAL: NCT00000709
Title: An Open Trial of Zidovudine (AZT) Treatment of the AIDS Dementia Complex in Patients With AIDS or Low CD4+ Lymphocyte Counts
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 061; 11035 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: AIDS Dementia Complex; HIV Infections
Keywords: Neuropsychological Tests; AIDS Dementia Complex; Zidovudine; CD4-Positive T-Lymphocytes
MeSH Terms: conditions — AIDS Dementia Complex; HIV Infections | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To provide accurate and complete neurologic assessment of the course of the AIDS dementia complex in patients treated with zidovudine (AZT). The study will determine how frequently patients improve, how long improvement is sustained, and the magnitude and functional significance of improvement.

Individuals with AIDS frequently suffer central nervous system (CNS) problems that are characterized by cognitive, motor, and behavioral deficits, in a disorder known as AIDS dementia complex. Clinical experience suggests that its course is often progressive, going from initial symptoms to moderate or severe dementia within several months. Accumulating evidence now suggests that direct brain infection by the HIV virus is the likely cause of the AIDS dementia complex. Case reports suggest that therapy with AZT, which has been shown to be a strong inhibitor of HIV replication in vitro, may alleviate the AIDS dementia complex. This study will help define the natural history of the AIDS dementia complex in treated patients.

DETAILED DESCRIPTION:
Individuals with AIDS frequently suffer central nervous system (CNS) problems that are characterized by cognitive, motor, and behavioral deficits, in a disorder known as AIDS dementia complex. Clinical experience suggests that its course is often progressive, going from initial symptoms to moderate or severe dementia within several months. Accumulating evidence now suggests that direct brain infection by the HIV virus is the likely cause of the AIDS dementia complex. Case reports suggest that therapy with AZT, which has been shown to be a strong inhibitor of HIV replication in vitro, may alleviate the AIDS dementia complex. This study will help define the natural history of the AIDS dementia complex in treated patients.

All patients receive AZT for 24 weeks. Patients are seen weekly for the first 4 weeks, every other week for the next 8 weeks, and then every 4 weeks until the completion of the study for neuropsychological evaluation. This evaluation includes lumbar puncture, and either computerized tomography or magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylactic therapy for Pneumocystis carinii pneumonia (PCP); aerosol pentamidine is the preferred method.
* Maintenance anticonvulsant therapy following a seizure in the context of the AIDS dementia complex.
* Patients taking anticonvulsants should have their anticonvulsant blood levels measured prior to starting zidovudine (AZT) or with changes in AZT dosage.
* Phenytoin, carbamazepine, and valproic acid.
* Judicious use of benzodiazepams.
* For analgesia or fever, modest doses of aspirin, Tylenol, or ibuprofen.
* Use of major mood or central nervous system altering drugs is discouraged and should be documented.

Patients with the following are included:

* An estimated pre-illness IQ = or > 70.
* A general neurodiagnostic evaluation before entry which will include a computerized tomographic (CT) scan or magnetic resonance imaging (MRI) scan and a lumbar puncture.
* Stable or indolently progressive mucocutaneous Kaposi's sarcoma with < 25 lesions and onset of < 10 new lesions during the 30-day period prior to study entry.
* Chronic seizure disorders requiring anticonvulsant therapy as long as the seizures are not associated with a fixed neurologic deficit.
* A blood HIV culture and p24 antigen capture assay at the time of the lumbar puncture. A second p24 antigen assay on study entry. Informed consent form must be signed by the patient, legal guardian, or parent.

Active substance abuse that would limit a patient's cooperation or evaluation.

Exclusion Criteria

Co-existing Condition:

Patients with the following will be excluded from the study:

* Active, symptomatic AIDS-associated opportunistic infections requiring ongoing maintenance therapy.
* Persistent fever, active persistent diarrhea, or continued severe weight loss.
* Severe premorbid psychiatric illness.
* Confounding neurologic disease or deficit.
* Concurrent or previous central nervous system infections or neoplasms.
* Concurrent active neoplasms other than basal cell carcinoma of the skin and mucocutaneous Kaposi's sarcoma.

Concurrent Medication:

Excluded:

* Major psychotropic medication including tricyclic antidepressants, MAO inhibitors, phenothiazines, butyrophenones, barbiturates, or amphetamines.
* Cimetidine.
* Ranitidine.
* Probenecid.
* Indomethacin.
* Acyclovir (ACV) prophylaxis for recurrent Herpes simplex.

Patients with the following will be excluded from the study:

* Active, symptomatic AIDS-associated opportunistic infections requiring ongoing maintenance therapy.
* Persistent fever, active persistent diarrhea, or continued severe weight loss.
* Severe premorbid psychiatric illness.
* Confounding neurologic disease or deficit.
* Concurrent or previous central nervous system infections or neoplasms.
* Concurrent active neoplasms other than basal cell carcinoma of the skin and mucocutaneous Kaposi's sarcoma.

Prior Medication:

Excluded within 2 weeks of study entry or for greater than 2 weeks of therapy:

* Zidovudine (AZT).
* Patients must not have previously exhibited toxic reaction to AZT.
* Excluded within 30 days of study entry:
* Immunomodulators and biologic response modifiers, including systemic steroids.
* Any investigational agent.
* Cytotoxic chemotherapy for Kaposi's sarcoma.

Prior Treatment:

Excluded within 30 days of study entry:

* Radiation therapy.
* Excluded within 2 weeks of study entry:
* Blood transfusion.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50
Dates: Study Completion 1990-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: RW Price, Study Chair
Locations (12):
- United States (12):
  - UCLA CARE Ctr, Los Angeles, California
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington